CLINICAL TRIAL: NCT07060716
Title: GraftAssureDx Study: Validation of Donor-Derived Cell-Free DNA (Dd-cfDNA) for Kidney Transplant Monitoring
Brief Title: Validation of Donor-Derived Cell-Free DNA (Dd-cfDNA) for Kidney Transplant Monitoring
Status: Recruiting | Type: Observational
Sponsor: Insight Molecular Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-001
Record Dates: First submitted 2025-06-02; First posted 2025-07-11 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplant Rejection; Cell-free DNA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: donor-derived cell-free DNA test — A donor-derived cell-free DNA (dd-cfDNA) test used to measure the concentration of total cell-free DNA and the fractional abundance of the dd-cfDNA.

SUMMARY:
The goal of this observational study is to learn if the donor-derived cell-free DNA (dd-cfDNA) test can assess rejection in kidney transplant recipients. Participants will have blood and urine collected at their study visit.

Researchers will compare results of the GraftAssureDx to rejection detected by standard-of-care graft biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older
2. At least 12 calendar days have elapsed since the subject received a kidney transplant.
3. Subject has provided legally effective informed consent
4. Subject agrees to comply with all study procedures

Exclusion Criteria:

1. Kidney donor is an identical twin of the subject.
2. The subject has another previously transplanted organ in situ.
3. Subject has received a hematopoietic stem cell transplant.
4. Subject has received a bone marrow graft.
5. Subject has self-reported as pregnant.
6. In the opinion of the investigator, the subject's participation in the study would pose a risk to data integrity or to the subject's safety and welfare.

Sample Inclusion Criteria:

1. A graft biopsy is obtained within ±1 week of blood draw.

* If blood draw is obtained after biopsy, blood draw should be taken at least 2 days after an uncomplicated biopsy procedure.

Sample Exclusion Criteria:

1. Sample collected from someone that had an invasive graft biopsy ≤ 48 hours prior to blood draw.
2. Sample collected from subject that received immunosuppressive treatment for biopsy-proven acute rejection ≤ 30 days prior to blood draw
3. Sample collected from subject that received a blood transfusion ≤ 30 days prior to blood draw.
4. Sample collected from a subject that provided another sample for the study within the past 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have received a kidney transplant at centers in the United States and Germany will be invited to participate.
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical validation of the dd-cfDNA test when compared to biopsy-confirmed rejection | Samples tested after final assay cutoffs have been established will be analyzed to demonstrate clinical performance of the investigational assay. This testing will occur from enrollment to 18 weeks after acquisition of the samples.
  Relative percentage of dd-cfDNA levels of 0.5% and absolute values of 50cp/mL are considered to be the diagnostic cutoff for rejection, which will be refined during the first study phase.
Clinical validation of the dd-cfDNA test when compared to biopsy-confirmed rejection | Samples tested after the final assay cutoffs have been established will be analyzed to demonstrate clinical performance of the investigational assay. This testing will occur from enrollment to 24 weeks after acquisition of the samples.
  Clinical sensitivity of the dd-cfDNA test shall be better or equal to published values (≥56%). Current literature shows an average sensitivity of 69% with a SD of 13%. Therefore, 56% represents the lower boundary (average - 1SD) of the distribution of published values.
Clinical validation of the dd-cfDNA test when compared to biopsy-confirmed rejection | Samples tested after the assay final cutoffs have been established will be analyzed to demonstrate clinical performance of the investigational assay. This testing will occur from enrollment to 24 weeks after acquisition of the samples.
  Clinical Specificity of the dd-cfDNA test shall be better or equal to published values (≥75%). Current literature shows an average specificity of 81% with a SD of 6%. Therefore, 75% represents the lower boundary (average - 1SD) of the distribution of published values.
Clinical validation of the dd-cfDNA test when compared to biopsy-confirmed rejection | Samples tested after the final assay cutoffs have been established will be analyzed to demonstrate clinical performance of the investigational assay. This testing will occur from enrollment to 24 weeks after acquisition of the samples.
  Predictive values are mathematically derived from sensitivity and specificity using the Bayes' theorem. Therefore, success criteria are defined as the lower boundary of the current literature at any given a priori probability. E.g., for an a priori probability of 20%, the lower boundary for NPV is 85%.
Clinical validation of the dd-cfDNA test when compared to biopsy-confirmed rejection | Samples tested after the final assay cutoffs have been established will be analyzed to demonstrate clinical performance of the investigational assay. This testing will occur from enrollment to 24 weeks after acquisition of the samples.
  Predictive values are mathematically derived from sensitivity and specificity using the Bayes' theorem. Therefore, success criteria are defined as the lower boundary of the current literature at any given a priori probability. E.g., for an a priori probability of 20%, the lower boundary for Positive Predictive Value (PPV) is 49%.

SECONDARY OUTCOMES:
ROC-AUC of dd-cfDNA vs. biopsy-confirmed rejection. | This testing will occur from assay cutoff up to 24 weeks after acquisition of the samples.
  The second endpoint is for investigational use only and therefore has no predefined success criteria.
Correlation between GraftAssureDx results and traditional biomarkers of kidney rejection (creatinine, estimated glomerular filtration rate, blood urea nitrogen). | This testing will occur from assay cutoff up to 24 weeks after acquisition of the samples.
  The second endpoint is for investigational use only and therefore has no predefined success criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Schuetz, MD, PhD, Study Chair — Insight Molecular Diagnostics
Locations (10):
- United States (8):
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor, Scott & White Research Institute, Dallas, Texas
  - Intermountain Health, Murray, Utah
- Germany (2):
  - Institute of Immunology - Transplantation Immunology, Heidelberg, Baden-Wurttemberg
  - Charite Universitatsmedizin, Berlin

IPD SHARING:
Plan to Share IPD: Undecided
only IPD used in the results publication